CLINICAL TRIAL: NCT01531400
Title: Investigation of Pain and Anxiety During Electrodiagnostic Examination Using Self-selected Music
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, Yu-Cheng Pei, Principle Investigator (Attending physician and clinical assistant professor), Chang Gung Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: cgmhpmr001
Record Dates: First submitted 2012-01-29; First posted 2012-02-13 (Estimated); Last update posted 2012-03-20 (Estimated); Status verified 2012-03

CONDITIONS: Pain; Anxiety
MeSH Terms: conditions — Pain; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- music (Experimental): Investigators played self-selected background music in the music group
  Interventions: Other: self-selected music
- no music (control) (No Intervention): Investigators played no music in the music group

INTERVENTIONS:
Other: self-selected music — Investigators played self-selected background music in the music group
  Other Names: self-selected background music
  Arms: music

SUMMARY:
The investigators hypothesized that self-selected music played during electrodiagnosis is effective in relieving the discomfort caused by the procedures.

ELIGIBILITY:
Inclusion Criteria:

Investigators recruited volunteer patient participants from patients referred to the electrodiagnosis laboratory of Department of Physical Medicine and Rehabilitation in a medical center using convenient sampling.

The inclusion criterion is:

* adult patient with working diagnosis of possible neurological disorder and
* is referred for both nerve conduction study and needle electromyography

Exclusion Criteria:

The exclusion criteria are:

* conscious disturbances,
* cognitive impairment, or
* language dysfunction.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2002-12; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Pain (Visual Analogue Scale) | baseline and after needle electromyography, to measure the "change" of pain

SECONDARY OUTCOMES:
Anxiety, assessed by Linear Analogue Anxiety Scale (LAAS) | baseline and after electromyography

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Cheng Pei, MD PhD, Principal Investigator — Attending Physician
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan, Taiwan